CLINICAL TRIAL: NCT03588065
Title: Health Education for Physiotherapy in Soccer Players
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped by insufficient funds
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, JORGE ENRIQUE MORENO COLLAZOS, Doctor Manual Therapy, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TERAPIA MANUAL
Record Dates: First submitted 2018-06-25; First posted 2018-07-17 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Soccer
Keywords: public health; Soccer
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: For the process of imparting health education strategies in face-to-face (conference) and ICT-mediated mode, a 4-week time was estimated where 4 educational sessions were held at a rate of one each week, lasting about 40 minutes, for part of two physiotherapists experts in the theme of injury prevention around the conceptual elements of human body movement, warm-up phases, postural hygiene, sports hygiene, nutrition and clothing. Interventions were carried out simultaneously in both groups of the study, so that one researcher taught the lecture modality in person (conference group), and the other supervised the participants while using the computers of the sports training institution.
Who Masked: Participant, Investigator
Masking Description: The FMS as a diagnostic evaluation test was applied in two moments with three blind physiotherapeutic evaluators with specialization in therapeutic physical activity and master in Physical Activity and Sports, with an experience of more than 5 years in the field of assessment of sport condition and clinical experience. in sport over 6 years in sports clubs in the region.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- attend education for TICS (Experimental): The educational activities were directed to soccer players belonging to Equidad, Bogotá-Colombia. Computerized media were used within the reach of footballers, applied with professionals of physical activity sciences under blind study methodology, using the new tendencies of Information and Communication Technologies (ICT) in Health Education. The investigators counted on the advice of the group manager of knowledge of the secretary of the district of the city of Bogotá. In the educational intervention seven aspects were addressed, distributed in four weekly modules for a total of four months
  Interventions: Diagnostic Test: FMS; Other: TICS
- attend education for conference (Active Comparator): The intervention arm descriptionTHE CONFERENCE include face-to-face sessions focused on the four aspects mentioned above for ICT. To this end, the theoretical elements of the concepts under study were taken into account: human body movement, warm-up phases, postural hygiene, sports hygiene, nutrition and clothing.
  The face-to-face sessions focused on the four aspects mentioned above for ICT. To this end, the theoretical elements of the concepts under study were taken into account: human body movement, warm-up phases, postural hygiene, sports hygiene, nutrition and clothing.
  Interventions: Diagnostic Test: FMS; Other: CONFERENCE
- attend for FMS (Sham Comparator): The FMS test was applied in two moments with three blind evaluators physiotherapists with specialization in therapeutic physical activity and master in Physical Activity and Sports, with an experience of more than 5 years in the field of assessment of sport condition and clinical experience in sport greater than 6 years in sports clubs in the region.
  Interventions: Diagnostic Test: FMS

INTERVENTIONS:
Diagnostic Test: FMS — The evaluation of the risk of sports injury was obtained from the score in the Functional Movement Screen test suite.
  The Functional Movement Screen (FMS) is a battery of tests that allows the integral assessment of the risk of injury, evaluating the basic patterns of movement and motor control through the performance of seven tests in which the combination of force is reflected muscle, flexibility, range of motion range, coordination, balance and proprioception
Other: TICS — The educational activities were directed to soccer players belonging to Equidad, Bogotá-Colombia. Computerized media were used within the reach of footballers, applied with professionals of physical activity sciences under blind study methodology, using the new tendencies of Information and Communication Technologies (ICT) in Health Education. The investigators counted on the advice of the group manager of knowledge of the secretary of the district of the city of Bogotá. In the educational intervention seven aspects were addressed, distributed in four weekly modules for a total of four months
  Arms: attend education for TICS
Other: CONFERENCE — The face-to-face educational intervention (conference) consisted of four educational sessions, distributed over four weeks during the sports transition period of the Equity sub-20 team. During these sessions, workshops (conferences) were held with the players following a face-to-face methodology . All these activities were concerted with the multidisciplinary team of the Equity football team and were carried out by the researcher at the University of La Sabana, a physiotherapist, who was studying the needs of the prevention of musculoskeletal injuries in football.
  Arms: attend education for conference

SUMMARY:
INTRODUCTION. Health education based on interventions with new information and communication technologies.

OBJECTIVE. To compare the effectiveness of an educational physiotherapy intervention in footballers, in face-to-face mode (conference) versus an intervention mediated by ICT, on the risk of medical injury with the Functional Movement Screen [FMS].

MATERIAL AND METHODS. A randomized clinical trial (RCT) was carried out. The population consisted of 100 participants divided into two groups (ICT n = 50) and (Conference n = 50), with an average age of 18.2 versus 18.3 years for a conference. and ICT respectively.

DETAILED DESCRIPTION:
Recruitment phase: In this phase the athletes were contacted to explain the objectives of the study and the interventions; those who agreed to participate filled out the questionnaire to verify the inclusion and exclusion criteria, later those who met the criteria gave written informed consent. This phase was held in a week in the sports team club Initial evaluation phase: In this phase, the contact form and the general characteristics of the population were filled out and the initial evaluation of knowledge about sports injuries was done in all the participants of the investigation. Likewise, the participants were assigned to each of the two interventions at random. For the random assignment, the Excel 2010® program was used, where random numbers were assigned to the sampling frame.

Intervention phase: The educational intervention in health was developed from physiotherapy in each of the groups (conference or mediated by ICT) according to the allocation group as explained below.

Final evaluation phase: The final evaluation of knowledge about the prevention of injuries in football was made to both groups of the investigation.

ELIGIBILITY:
Inclusion Criteria:

* Athletes over 18 years of age belonging to the La Equidad sports club.
* Athletes with a previous sporting age of more than three years.Athletes who have taken the entrance exam for the interdisciplinary team of the previous or initial physical condition of the La Equidad sports club.
* Resident in Bogotá or municipalities of Cundinamarca.

Exclusion Criteria:

* Alterations of perception or behavior that hinder educational interventions.
* Other co-morbidities reported by the user or in the clinical history of the sport that limit the intervention (Example: hearing loss, kyphosis, memory deficit or cognitive attention, visual limitation).
* Users who do not have training in educational computer skills.
* Not having a computer with an internet connection.

Ages: 18 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — SPORTS SELECTION SUB20
Enrollment: 100 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2017-10-08 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
SELF-AWARENESS QUESTIONNAIRE ON SPORTS INJURIES | 4 months
  A total of 17 questions were established, divided into seven categories of knowledge on the prevention of injuries, which should be addressed in the health education plan from Physiotherapy. The score was calculated as follows: each question answered correctly with the option of YES and NO had a point, the sum of the correct questions was made and divided by the number of questions. Using a rule of three this score was converted to a scale of 0 to 100.

SECONDARY OUTCOMES:
FMS | 4 months
  The scores of the seven movement patterns. If the athlete is able to make the movements without any compensation, receive a score of 3. If the athlete performs the movement with one or more compensations or with a difficulty to receive a score of 2. If the athlete is unable to reproduce the requested movement, receive a score of 1. If during the performance of the test the athlete presents pain, receive a score of zero and should be referred to a specialist. The maximum score for the sum of all movements is 21.

CONTACTS AND LOCATIONS:
Overall Officials: JORGE MORENO COLLAZOS, PHD, Principal Investigator — universidad cardenal herrera
Locations (1):
- Equidad Sport, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
does not apply